CLINICAL TRIAL: NCT06555055
Title: Trochlear Thickness and Its Effect on the Outcomes of Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Ibrahim barsoum (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, Ibrahim barsoum, Ass. lecturer., Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: Trochlear thickness in TKA
Record Dates: First submitted 2024-07-14; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; patellofemoral; TKA; Trochlear thickness
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- trochlear thickness change: Radiological Assessment of trochlear thickness of PFJ in primary TKR by preoperative and postoperative CT scan. and observing Effects of Ct Different measures changes in trochlear thickness on short term TKR outcomes
  Interventions: Other: CT trochlear thickness change

INTERVENTIONS:
Other: CT trochlear thickness change — Preoperative and postoperative CT scan measuring trochlear thickness of PFJ was defined as distance from deepest part of trochlea and line tangential to the anterior aspect of the femoral cortex. It was assessed on the sagittal cuts.
  CT images will be viewed using Sante DICOM viewer version 5.4.2 and image fusion will be done using Overlay multiple image software.
  Two observers will measure the angles and the intraobserver and interobserver reliabilities will be assessed for consistency by the intraclass correlation coefficient (ICC) and reliability coefficient using the SPSS software

SUMMARY:
Total knee arthroplasty (TKA ) is the gold standard treatment for advanced knee osteoarthritis. only 85% (75% to 92%) of patients with total knee arthroplasty are satisfied with their operations and 30% develops patellofemoral complications.

Numerous biomechanical studies suggest that patellofemoral tracking is not always restored to physiological values, because the prosthetic trochlea may differ from the native trochlea. no study has been con-ducted to investigate the thickness of the trochlear groove and its effect on the outcome of Total knee replacement (TKR), So many people has different measurements of trochlear thickness which may affect Patellofemoral joint (PFJ) so knowing of native trochlear thickness in patients with KNEE Osteoarthritis (OA) can affect the outcomes of total knee arthroplasty.

DETAILED DESCRIPTION:
Total knee arthroplasty is the gold standard treatment for advanced knee osteoarthritis. In spite of the great advance in the prosthesis design, surgical techniques and rehabilitation programs, only 85% (75% to 92%) of patients with total knee arthroplasty are satisfied with their operations and 30% develops patellofemoral complications. Patellofemoral complications after TKR are usually caused by multiple factors related to surgical technique (e.g., implant positioning and sizing, soft-tissue balancing, patellar resurfacing, etc.) and implant design (e.g., trochlear thickness, sagittal curvature, patellar component shape).

Numerous biomechanical studies suggest that patellofemoral tracking is not always restored to physiological values, because the prosthetic trochlea may differ from the native trochlea.

Theoretically decreasing of contact area distance of trochlea might increase the contact pressure in the patellofemoral joint. The increased contact pressure will elevate the stress in the subchondral bone of the patellofemoral joint, which is hypothesized to be a cause of patellofemoral pain.

A mechanical experiment was performed in an attempt to analyze the influence of thickening of the patella on the knee extension movement. The measurement show that anterior advancement of the extensor apparatus at the level of the patella gives a mechanical advantage, enabling the quadriceps to extend the knee with the use of less force. so increase thickness of patella affects the quadriceps function but no study has been shown the effect of trochlear thickness on quadriceps or patellofemoral joint.

Nonetheless, no study has been con-ducted to investigate the thickness of the trochlear groove and its effect on the outcome of TKR, So many people has different measurements of trochlear thickness which may affect PFJ so knowing of native trochlear thickness in patients with KNEE OA can affect the outcomes of total knee arthroplasty.

Preoperative and postoperative radiography (CT scan) can provide an adequate measurement of trochlear thickness which will help in understanding more about PFJ and its effect in the total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* Advanced knee osteoarthritis in which total knee arthroplasty is indicated

Exclusion Criteria:

* Revision total knee arthroplasty
* Previous osteotomy around the knee
* Post traumatic knee arthritis
* Inflammatory knee arthritis

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with primary knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Functional outcome | preoperative and six months postoperatively
  knee society score (KSS).
Functional Outcome | preoperative and six months postoperatively
  Patellofemoral score (Barlett patellofemoral score).
Functional Outcome | preoperative and six months postoperatively
  ROM

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim B Anis, MS, Principal Investigator — Ain Shams University; Wael S Abd El Mageed, MD, Study Director — Ain Shams University; Sherif M El Sayed, MD, Study Director — Ain Shams University; Zeiad M Zakaria, MD, Study Director — Ain Shams University; Mohmed E Awad, MD, Study Director — Ain Shams University
Locations (1):
- Ain Sahms University, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ranawat CS, Flynn WF Jr, Saddler S, Hansraj KK, Maynard MJ. Long-term results of the total condylar knee arthroplasty. A 15-year survivorship study. Clin Orthop Relat Res. 1993 Jan;(286):94-102. PMID 8425373
- [Result] Healy WL, Wasilewski SA, Takei R, Oberlander M. Patellofemoral complications following total knee arthroplasty. Correlation with implant design and patient risk factors. J Arthroplasty. 1995 Apr;10(2):197-201. doi: 10.1016/s0883-5403(05)80127-5. PMID 7798101
- [Result] Dejour H, Walch G, Neyret P, Adeleine P. [Dysplasia of the femoral trochlea]. Rev Chir Orthop Reparatrice Appar Mot. 1990;76(1):45-54. French. PMID 2140459